CLINICAL TRIAL: NCT04662424
Title: Effect of Music in Labor in Women Who Underwent Induction of Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 301/20
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MUSIC (Experimental): music in labor
  Interventions: Other: music in labor
- control (No Intervention): no music during labor

INTERVENTIONS:
Other: music in labor — Women in the intervention group will be offered music in labor, defined listening to music from the randomization until the delivery of the baby. Women had the possibility to select the songs at their discretion
  Arms: MUSIC

SUMMARY:
Women's experience of pain during labor varies greatly, and pain control is a major concern for obstetricians. Several methods have been studied for pain management for women in labor, including drug and non-drug interventions Most methods of non-pharmacological pain management are non-invasive and appear to be safe for mother and baby, including immersion in water, relaxation, acupuncture, and massage. However, their efficacy is unclear, and based mostly on non-randomized studies. On the other hand, there are strong data to support the efficacy of pharmacological methods, including epidural analgesia, which improves pain relief but increase the incidence of operative vaginal delivery Recently a clinical trial showed that music in labor was associated with maternal benefits in women who underwent spontaneous vaginal delivery. However, the effect of music in labor in women undergoing induction of labor is still a subject of debate.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Singleton gestation
* Vertex presentation
* Induction of labor, i.e. cervical ripening with prostaglandins
* Gestational age between 37 and 42 weeks

Exclusion Criteria:

* Multiparous womne
* Multiple gestations
* Preterm labor
* Preterm premature rupture of membranes
* Induction of labor with oxytocin and without prostaglandins
* Induction of labor with balloon
* High risk pregnancies, including hypertensive disorders of pregnancies, diabetes, intrauterine growth restriction, fetal abnormalities.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 30 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-02-20 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
mean pain level during the active phase of labor | at the time of the active phase of labor
  assessed by Visual Analog Scale (VAS) for Pain

SECONDARY OUTCOMES:
Mean anxiety level during the active phase of labor, second stage, and at post-partum | at the time of the active phase of labor
  assessed by Visual Analog Scale (VAS) for anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Saccone, MD, Principal Investigator — Federico II University
Locations (1):
- Gabriele Saccone, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided
unplanned